CLINICAL TRIAL: NCT00977587
Title: Effect of Saccharomyces Cerevisiae CNCM I-3856 on Faecal Proteases and Symptoms Associated With IBS-D and Postinfective Bowel Dysfunction
Brief Title: Saccharomyces Cerevisiae CNCM I-3856 Treatment in Irritable Bowel Syndrome With Diarrhea (IBS-D) and Post Infective Bowel Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to get MHRA approval for formulation in present form
Sponsor: University of Nottingham (Other)
Collaborators: Lesaffre International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09075
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2012-01

CONDITIONS: Irritable Bowel Syndrome; Post Infective Bowel Dysfunction
Keywords: irritable bowel syndrome; faecal serine proteases
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saccharomyces Cerevisiae CNCM I-3856 (Active Comparator): 2 weeks of treatment with Saccharomyces Cerevisiae CNCM I-3856 1 capsule twice a day, 500 mg per capsule (5 X109 living cells). Living cells are estimated by the method of colony forming units (cfu).
  Interventions: Drug: Saccharomyces Cerevisiae CNCM I-3856
- placebo (Placebo Comparator): Capsules will contain 500 mg of the following formulation and will not contain Saccharomyces cerevisiae CNCM I-3856:
  * Calcium phosphate, Dibasic 472.0 mg
  * Maltodextrin DE14 112.1 mg
  * Vegetal magnesium stearate 5.9 mg subjects will take one capsule twice a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Saccharomyces Cerevisiae CNCM I-3856 — Saccharomyces cerevisiae CNCM I-3856, 500 mg per capsule (5 X109 living cells). Living cells are estimated by the method of colony forming units (cfu).subjects will take 1 capsule twice a day
  Arms: Saccharomyces Cerevisiae CNCM I-3856
Drug: placebo — Placebo: Capsules will contain 500 mg of the following formulation and will not contain Saccharomyces cerevisiae CNCM I-3856:
  * Calcium phosphate, Dibasic 472.0 mg
  * Maltodextrin DE14 112.1 mg
  * Vegetal magnesium stearate 5.9 mg subjects will take one capsule twice a day
  Arms: placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common condition characterised by abdominal pain or discomfort and altered bowel habit affecting up to 10% of the population. There are several groups of patients that are based on differing bowel patterns including IBS with diarrhea (IBS-D) and those with post infective IBS (PI-IBS) whose symptoms begin after an acute infection. Saccharomyces cerevisiae, the yeast used in bread making has been shown to reduce the duration of infectious diarrhoea. Part of the benefit maybe that it can destroy bacterial toxins. Recent studies suggest an increase in proteases (chemicals which breakdown proteins) in the stool of patients with IBS-D. The investigators think that this yeast may benefit patients with IBS-D and PI-IBS by reducing the amount of protease in stool. This is important because proteases have been shown to be potentially important in generating some of the discomfort experienced by patients. The investigators will study patients with chronic IBS-D who will receive 2 weeks treatment with the yeast or placebo followed by a 4 week gap and then a further 2 week treatment with placebo or the yeast, with the treatments allocated randomly. The investigators will also study 30 subjects who still have persistent loose bowel function 6 weeks after an infection with Campylobacter jejuni, one of the commonest causes of gastroenteritis in the UK. Subjects will be randomised to take either the yeast or placebo for 4 weeks . In both studies, the investigators will examine the effect of treatment on stool proteases, stool frequency and consistency and abdominal discomfort; the investigators will also take blood samples to examine some aspects of immune system function. The results of the study may suggest how yeast provides a benefit in patients with IBS and diarrhea and will provide data for a larger clinical trial.

DETAILED DESCRIPTION:
The participant involvement in study 1 & 2 will last 15 & 9 weeks respectively. Study1 has a cross over design so each participant will receive two 2 week treatment periods (1 of placebo and 1 of active) with a 4 week washout period in between. The order with which they receive the treatment will be decided randomly. The study starts with a screening period lasting 1 week. If, at the end of screening, they are still eligible they will be enrolled and start randomised treatment. Once the participant has received both treatments the study finishes.

Study 2 is a parallel group design. Subjects who submit a stool sample which proves to be positive for Campylobacter will be sent an invitation to take part. All subjects will be asked to complete a bowel symptom questionnaire and attend to provide a stool sample (enrolment visit). A blood sample will be taken at this visit.

After a further 4 weeks subjects will attend again, bringing with them a stool sample and stool symptom diaries. A blood sample will be taken. At this time, if they are still symptomatic they will be invited to take part in the randomised placebo controlled trial taking yeast or placebo for 5 weeks, after which they will again attend with stool diaries and provide a final stool and blood sample. The blood sample will be used to see, if antibodies to C. jejuni antigens predicts recovery and whether this is altered by yeast treatment. Those that are asymptomatic will not take part in the RCT but will return at 9 weeks with a further stool and blood sample.

We will also invite 15 healthy volunteers, free from gastrointestinal complaints to attend on 3 occasions mimicking visits 1-3 by providing stool and blood samples so we can define the normal variability in stool composition in health. As with the other subjects they will be required to avoid antibiotics and probiotics during the study.

End of Studies The last visit of the last subject.

SELECTION AND WITHDRAWAL OF PARTICIPANTS Recruitment Study 1 Participants for study 1 will be recruited from Professor Spiller's patients who have previously taken part in research studies and have indicated that they would like to be contacted about future relevant research projects. This secure password protected database is held within the Nottingham Digestive Diseases Centre and contains patient's names and addresses to allow mailing of invitation letter.

The investigator or their nominee, i.e. a member of the participant's usual care team, will make the initial approach to the patient by letter to the patient using a ethically approved invitation letter enclosing a copy of the information sheet and inform the participant of all aspects pertaining to participation in the study.

Study 2 Currently all patients who submit a stool sample positive for C jejuni to the Public Health laboratory receive a letter form Professor Neal asking for details about eating out and pet's illnesses as part of routine surveillance. This letter will have an information sheet enclosed and an invitation to take part in Study 2 We will also recruit 15 healthy volunteers who have responded to an advert displayed on public notice boards at University Hospital Nottingham. On responding, they will then be sent an information sheet and details of the study and who to contact if they are interested in taking part.

ELIGIBILITY:
Inclusion Criteria:

Study 1 and 2:

* Male or female aged 18-75 years
* Subjects who are able to give informed consent

Study 1:

* IBS-D patients meeting Rome III Criteria

Study 2:

* Subjects with stool cultures positive for Campylobacter jejuni
* Healthy volunteer controls

Exclusion Criteria:

* Subjects that, in the opinion of the investigator, are considered unsuitable.
* Subjects who have had abdominal surgery which may cause bowel symptoms similar to IBS (Please note, appendicectomy and cholecystectomy is not an exclusion).
* Subjects with a known intolerance to yeast.
* Subjects taking immunosuppressant medication, e.g. long term steroids, or who might otherwise be immunocompromised.
* Subjects who have had a recent course of antibiotics (in the last 28 days).
* Subjects unable to stop anti-diarrhoeal drugs.
* Subjects currently participating in another clinical trial or who have been in a trial in the previous three months.
* Patients with known gastrointestinal diseases including coeliac disease and inflammatory bowel disease.
* Regular consumption of drugs known to alter bowel habit (see concomitant medication).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Change in faecal serine protease activity | at 4 and 9 weeks for study 1 and 10 weeks for study 2

SECONDARY OUTCOMES:
Stool consistency | at 4 and 9 weeks for study 1 and ten weeks for study 2
Stool frequency | at 4 and 9 weeks for study 1 and 10 weeks for study 2
Number of mucus septae per high power filed | at 4 and 9 weeks for study 1 and 10 weeks for study 2
In vitro effect of Saccharomyces cerevisiae CNCM I-3856 supernatant on IBS-D faecal proteases | at week one for both studies
Bacterial diversity assessed by similarity indices | at week 1 for both studies at week 4 and 9 for study 1 and week 10 for study 2

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MB B Chir Cantab, MSc Lond, MD, Principal Investigator — Nottingham Digestive Diseases Centre and Biomedical Research Unit
Locations (1):
- Nottingham University Hospital, Nottingham, Nottinghamshire, United Kingdom